CLINICAL TRIAL: NCT04154995
Title: Long-term Recovery of Patients Admitted to the Intensive Care Unit
Brief Title: Intensive Care Unit Recovery
Acronym: ICU-RE
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Dr., Frisius Medisch Centrum
Other Study IDs: RTPO 1055
Record Dates: First submitted 2019-05-20; First posted 2019-11-07 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Post Intensive Care Unit Syndrome; Intensive Care Unit Acquired Weakness; Critical Illness
Keywords: Long-term recovery; Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term ICU patients: Patients with a ICU length of stay of at least 48 hours.
  Interventions: Diagnostic Test: Venipuncture; Diagnostic Test: Ultrasound Quadriceps Muscles

INTERVENTIONS:
Diagnostic Test: Venipuncture — Blood testing at 3, 6 and 12 months
Diagnostic Test: Ultrasound Quadriceps Muscles — Ultrasound measurement of quadriceps muscle mass and health

SUMMARY:
Survival rates of patients with critical illness have increased due to improved facilities and treatment methods in the intensive care unit (ICU). Despite surviving critical illness, patients often face a difficult road of rehabilitation after discharge from the ICU or the hospital ward. A large body of evidence indicates that critical illness survivors suffer from physical and mental health problems, reflected in a reduced health related quality of life. However, detailed studies on longer-term outcomes and physical and mental recovery are lacking. In order to develop a tailored aftercare intervention program for critical care survivors a detailed description of the specific health problems is necessary. The aim of this study is to evaluate the change in health-related quality of life (HRQoL) and physical and mental health of critical illness survivors.

DETAILED DESCRIPTION:
Introduction

Survival rates of patients with critical illness have increased due to improved facilities and treatment methods in the intensive care unit (ICU). Despite surviving critical illness, patients often face a difficult road of rehabilitation after discharge from the ICU or the hospital ward. A large body of evidence indicates that critical illness survivors suffer from physical and mental health problems, reflected in a reduced health related quality of life. However, detailed studies on longer-term outcomes and physical and mental recovery are lacking. In order to develop a tailored aftercare intervention program for critical care survivors a detailed description of the specific health problems is necessary. The aim of this study is to evaluate the change in health-related quality of life (HRQoL) and physical and mental health of critical illness survivors.

Methods

In this prospective single-center observational study 80 long-term ICU-patients will be included within six months. In addition to standard ICU care, the following measurements will be taken within 72 hours after ICU-admission: ultrasound measurements of the quadriceps, bioimpedance, plasma glutamine concentration and HRQoL using the RAND-36 item Health Survey (RAND-36). If the patient is unable to fill in the questionnaire, a proxy will be asked for this. The ultrasound, bioimpedance and plasma glutamine measurements will be repeated weekly in case the patient remains in ICU. When the patient is able to perform physical tests, hand grip strength and Morton Mobility Index measurements will be conducted weekly. After ICU-discharge, patients will be contacted by phone after 1,5, 4,5 and 9 months for an interview about dietary - and exercise habits. Furthermore, patients visit the specialised outpatient ICU clinic at 3, 6 and 12 months after ICU-discharge. Before this visit, patients will be asked to fill in a combination of questionnaires regarding mental health and HRQoL, specifically the RAND-36, the Hospital Anxiety and Depression Scale, the Short Fatigue Questionnaire, the Coping Inventory for Stressful Situations, the Trauma Screening Questionnaire, the Cognitive Failure Questionnaire and the Happiness Index. Secondly, blood samples are taken to measure c-reactive protein, hemoglobin, creatinine, albumin, glucose, glutamine, and biomarkers for mitochondrial dysfunction. Also, the following physical measures will be taken: bioimpedance measures, ultrasound of the quadriceps, hand grip strength, Morton Mobility Index, Barthel Index Score, Berg Balance Scale and the 6 minute walking test with pulse oximetry.

Statistical analysis Variables will be summarised as, mean±standard deviation (SD), median [interquartile range, IQR] and number (percentage) for continuous or categorical variables, respectively.

RAND-36 measures will be used to establish non-recovery patient groups. If appropriate, multivariate analyses will be conducted to identify risk factors with prognostic value for 1 year post-ICU recovery. Significance levels will be set at p<0.05 for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Expected length of stay ICU ≥ 48 hours

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU with an expected stay of 48 hours or longer will be asked for consent to participation of this study. The average number of patients admitted per year to the ICU of Medical Centre Leeuwarden with a length of stay (LOS) > 48 hours is 230. Due to practical limitations, we aim to include a maximum number of 80 patients within a six-month period. After six months, the inclusion will be stopped irrespective of the number of included patients.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life | Baseline, 3, 6 and 12 months
  Change in HRQoL using the Dutch translation of the Research and Development-36 item Health Survey (RAND-36). This survey consists of nine subscales (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health perception and health change). Total subscale scores are reported with a range of 0 to 100 percent. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Quadriceps muscle layer thickness | Baseline, 3, 6 and 12 months
  Quadriceps ultrasound thickness measured in mm. Values below reference values indicate a worse outcome.
Bioimpedance measurement in BIVA | Baseline, 3, 6 and 12 months
  Bioimpedance measurements (baseline from standard care clinical data) measured using bioelectrical impedance vector analysis. Phase angle (degrees), reactance (Ohm) and resistance (Ohm) are measured. Fat free mass (kg) and total body water (l) are calculated using these measurements. Values above or below reference values indicate a worse outcome.
Hand grip strength | Baseline, 3, 6 and 12 months
  Hand grip strength test of the left and right hand in kg. Values below reference values indicate a worse outcome.
Walking distance | 3, 6 and 12 months
  6-minute walk test measures are taken in meters. Values below reference values indicate a worse outcome.
physical activity | Baseline, 3, 6 and 12 months
  Morton Mobility Index scores are taken. This survey/physical test questionnaire consists of 15 questions with a scoring range of 0-19. A lower score indicates a worse outcome.
Blood c-reactive protein concentration | Baseline, 3, 6 and 12 months
  C-reactive protein (baseline from standard care clinical data) levels from blood samples in mg/L. Higher values indicate a worse outcome.
Blood creatinine concentration | Baseline, 3, 6 and 12 months
  Creatinine (baseline from standard care clinical data) levels from blood samples in μmol/L. Values below or above reference values indicate a worse outcome.
Blood haemoglobin concentration | Baseline, 3, 6 and 12 months
  Haemoglobin (baseline from standard care clinical data) levels from blood samples in mmol/L. Values below or above reference values indicate a worse outcome.
Blood albumin concentration | Baseline, 3, 6 and 12 months
  Albumin (baseline from standard care clinical data) levels from blood samples in g/L. Values below or above reference values indicate a worse outcome.
Blood glucose concentration | Baseline, 3, 6 and 12 months
  Glucose non fasting (baseline from standard care clinical data) from blood samples in mmol/l. Values below or above reference values indicate a worse outcome.
Blood glutamine concentration | Baseline, 3, 6 and 12 months
  Glutamine levels from blood samples in mmol/l. Values below reference values indicate a worse outcome.
Biomarkers for mitochondrial dysfunction | Baseline, 3, 6 and 12 months
  Levels of biomarkers for mitochondrial dysfunction from blood samples.
Fatigue | 3, 6 and 12 months
  Change in subjective fatigue using the Dutch short-fatigue questionnaire/Verkorte Vermoeidheidsvragenlijst (VVV). This survey consists of 4 questions and has a total scoring range of 7-24 in which a lower score indicates a worse outcome.
Depression | 3, 6 and 12 months
  Change in mental health using the Hospital anxiety and depression scale (HADS). This survey consists of two subscales with seven questions each. The score range is 0-21 for each subscale in which a higher score indicates a worse outcome.
  * Coping inventory for stressful situations (CISS-21)
  * Trauma screening questionnaire (TSQ)
  * Happiness Index (HI)
  * Cognitive functioning questionnaire (CFQ-25)
Coping with stressful situations | 3, 6 and 12 months
  Identification of coping style using the Coping inventory for stressful situations (CISS-21). This survey consists of three subscales with 7 questions each. The score range is 7-30 for each subscale. The subscale with the highest score is indicated as the most prominent coping style at that moment.
Trauma | 3, 6 and 12 months
  Change in trauma symptoms using the trauma screening questionnaire (TSQ). This survey consists of 10 questions with a total score range of 0-10 in which a higher score indicates a worse outcome.
Subjective Happiness | 3, 6 and 12 months
  Subjective happiness is assessed using the Happiness Index (HI). This questionnaire consists of one question with a score range of 0-10. A lower score indicates a worse outcome.
Cognitive functioning | 3, 6 and 12 months
  Change in cognitive functioning is evaluated using the Cognitive failure questionnaire (CFQ-25). This survey consists of 25 questions with a total score range of 25-125. A higher score indicates a worse outcome.
Changes in dietary and exercise pattern | 1,5, 4,5 and 9 months
  Dietary and exercise patterns are assessed using a 24-hour diet and exercise recall interview. The participant is asked to recall all food intake and exercise of the day before. The interviewer makes a written report of the details and compares the intake and exercise to reference values.

OTHER OUTCOMES:
Baseline demographic data | Baseline, 3, 6 and 12 months
  Age (yr), gender (male/female/other), height (cm), weight (kg), weight before ICU admission (kg), weight change (kg), health care utilization (average number of visits to a health care professional a month), living situation (number of household members), and work situation (paid job/volunteering job/no job + hours).
Clinical data during ICU stay from standard care | Retrieved at 12 months from electronic patient data file
  Standard care ICU-characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided